CLINICAL TRIAL: NCT06472323
Title: The Efficacy and Safety of Pulsed Radiofrequency(PRF) Combined With Platelet-rich Plasma Versus PRF Alone for the Trigeminal Neuralgia
Brief Title: The Efficacy and Safety of Pulsed Radiofrequency Combined With Platelet-rich Plasma for the Trigeminal Neuralgia
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management Affiliation: Beijing Tiantan Hospital, Beijing Tiantan Hospital
Other Study IDs: KY2023-263-03-1
Record Dates: First submitted 2024-06-10; First posted 2024-06-25 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Trigeminal Neuralgia, Idiopathic; PRP
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRF+PRP: The puncture point was located 3cm outside the corners of the mouth of the affected side, using the Hartel technique. Under CT guidance, the trocar then was inserted through the ipsilateral foramen ovale to the Gasserian ganglion. After accurately puncturing the foramen ovalis, remove the cannula needle core and connected with RF electrode (PMK-21-100, Baylis, Canada) and the RF generator. Electrical stimulation was carried out at 50 Hz to determine the sensory threshold and at 2 Hz to determine the motor threshold. The RF generator was set to the manual PRF mode with a standard setting of 42°C, the UP knob was turned to increase the output voltage until the maximum voltage (bearable without causing pain in conscious patients)was reached; 120 s, 2 times. After removing the RF electrode in the combined treatment group, 2 ml of LP-PRP mixture was injected slowly into the Gasserian ganglion and mandibular nerve.
  Interventions: Procedure: PRF+PRP, PRF
- PRF: The puncture point was located 3cm outside the corners of the mouth of the affected side, using the Hartel technique. Under CT guidance, the trocar then was inserted through the ipsilateral foramen ovale to the Gasserian ganglion. After accurately puncturing the foramen ovalis, remove the cannula needle core and connected with RF electrode (PMK-21-100, Baylis, Canada) and the RF generator. Electrical stimulation was carried out at 50 Hz to determine the sensory threshold and at 2 Hz to determine the motor threshold. The RF generator was set to the manual PRF mode with a standard setting of 42°C, the UP knob was turned to increase the output voltage until the maximum voltage (bearable without causing pain in conscious patients)was reached; 120 s, 2 times.
  Interventions: Procedure: PRF+PRP, PRF

INTERVENTIONS:
Procedure: PRF+PRP, PRF — Under CT guidance, the trocar then was inserted through the ipsilateral foramen ovale to the Gasserian ganglion of the patient. After puncturing the foramen ovalis, remove the cannula needle core and connected with RF electrode (PMK-21-100, Baylis, Canada) and the RF generator. Electrical stimulation was carried out at 50 Hz to determine the sensory threshold and at 2 Hz to determine the motor threshold. The RF generator was set to the manual PRF mode with a standard setting of 42°C, the UP knob was turned to increase the output voltage until the maximum voltage (bearable without causing pain in conscious patients)was reached; 120 s, 2 times. After removing the RF electrode in the combined treatment group, 2ml of LP-PRP mixture was injected slowly into the Gasserian ganglion and mandibular nerve and PRF group only receive PRF treatment.

SUMMARY:
Trigeminal neuralgia (TN), characterized by brief, recurrent paroxysms of lancinating pain in the distribution of 1 or more branches of the trigeminal nerve (fifth cranial nerve [CNV]), is one of the most common, severe forms of neuropathic pain. Current standard of care for TN is the sodium channel blockers such as carbamazepine or oxcarbazepine. Surgical treatments involve percutaneous procedures, stereotactic radiosurgery and open surgical treatment. Each of these treatments have drawback. In recent years, pulsed radiofrequency (PRF) has been shown to be a promising treatment option for TN. But it was reported that the long-term outcomes of PRF was not satisfactory. Thus, there is an overwhelming need for finding a safe, nondestructive treatment option that is more effective for TN. PRP releases a variety of bioactive factors and adhesion proteins, which are responsible for activating hemostatic cascade reaction, synthesizing new connective tissue and vascular reconstruction, to initiate tissue repair processes. Autologous platelet-rich plasma (PRP) is the processed liquid fraction of autologous peripheral blood with a platelet concentration above the baseline. Studies have shown that it can reduce inflammation and promote nerve repair so it has also shown broad prospects in treating neuropathic pain. In 2012, Doss AX. published a case report indicated that PRP might be effective in TN treatment. In 2023, a randomized controlled study showed that CT-guided PRF combined with PRP can effectively treat postherpetic neuralgia (PHN), and the therapeutic effect is better than that of traditional PRF combined with glucocorticoid therapy in patients with PHN, which is similar to TN in pathology. Thus, we suppose that PRF combined with PRP might show better effectiveness than PRF alone for TN and conducted a prospective trail comparing the clinical efficacy and safety of PRP combined with PRF versus PRF alone. This study is designed as a prospective cohort study, open-label study with a 12 months follow-up period, to compare the efficacy of PRF combined with PRP versus PRP alone for TN treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of TN was established according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria (1).
2. Aged 18 to 75 years.
3. Had a score of at least 4 on a Numeric Rating Scale (NRS-11) (NRS; range, 0-10; higher scores indicate more severe pain) and could't be alleviated effectively by means of conservative medical therapy, such as carbamazepine, oxcarbazepine.
4. Agreed to sign the informed consent form.

Exclusion Criteria:

1. Patients presenting classic TN or secondary TN (i.e., multiple sclerosis).
2. Infection at the site of needle entry or systemic infecting.
3. A history of psychiatric disease.
4. Disorder indicated in the results of routine blood tests, hepatic function, renal function, coagulation function, electrocardiogram, or chest x-ray.
5. Serious systemic diseases such as uncontrolled hypertension or diabetes, and cardiac dysfunction (New York Heart Association grade II-III).
6. A history of abuse of narcotics.
7. A history of receiving CRF to the Gasserian ganglion or peripheral branches, glycerol rhizolysis, balloon compression, Gamma knife, or any other neuroablative treatments.
8. A history of receiving microvascular decompression.
9. Use of anticoagulants or antiplatelet agent, eg. acetylsalicylic acid.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main purpose of this study will be to compare the effectiveness of PRF combined with and without PRP, evaluated 1 year after the procedure. The effectiveness of PRF combined PRP group after 1 year is supposed to be 90%, and that of the high-voltage PRF group was 69% (29) (The α is 0.05, and the power is 90%). Power Analysis and Sample Size (PASS) V.15.0 software (NCSS Corporation, Kaysville, UT, USA) was used to compute the sample size. The results show that 73 patients will be required in each group. However, Accounting for 10% loss to follow-up and an additional 40% loss after propensity score matching, 135 patients will be recruited in each group. Therefore the total sample size of this study is supposed to be 270 participants.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The response rate of treatment | After 12 months
  Patients with BNI scores of I to III were considered to respond to treatment (Table 2).

SECONDARY OUTCOMES:
BNI scores | day 1; after 1 and 2 weeks; and after 1, 2, 3, 6, and 12 months following the procedure
  I No pain, off medications II Occasional pain, off medications IIIa No pain, continued use of medications IIIb Pain persists, but adequately controlled with medications IV Pain not adequately controlled with medications V No relief
The response rate of treatment | 1day, 1 and 2 weeks, 1, 2, 3, and 6 months following the procedure
  The response rate of treatment
Anticonvulsant consumption | After 1 day, 1 and 2 weeks, and after 1, 2, 3, 6, and 12 months following the procedure
  Dose of carbamazepine or oxcarbazepine
Scores on the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) | After 1, 3, 6, and 12 months following the procedure
  Scores on the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University in Beijing, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Ren H, Zhao C, Wang X, Shen Y, Meng L, Luo F. The Efficacy and Safety of the Application of Pulsed Radiofrequency, Combined With Low-Temperature Continuous Radiofrequency, to the Gasserian Ganglion for the Treatment of Primary Trigeminal Neuralgia: Study Protocol for a Prospective, Open-Label, Parall. Pain Physician. 2021 Jan;24(1):89-97. PMID 33400432
- [Background] Jia Y, Cheng H, Shrestha N, Ren H, Zhao C, Feng K, Luo F. Effectiveness and safety of high-voltage pulsed radiofrequency to treat patients with primary trigeminal neuralgia: a multicenter, randomized, double-blind, controlled study. J Headache Pain. 2023 Jul 18;24(1):91. doi: 10.1186/s10194-023-01629-7. PMID 37464283
- [Background] Luo F, Wang T, Shen Y, Meng L, Lu J, Ji N. High Voltage Pulsed Radiofrequency for the Treatment of Refractory Neuralgia of the Infraorbital Nerve: A Prospective Double-Blinded Randomized Controlled Study. Pain Physician. 2017 May;20(4):271-279. PMID 28535550
- [Background] Chong MS, Bahra A, Zakrzewska JM. Guidelines for the management of trigeminal neuralgia. Cleve Clin J Med. 2023 Jun 1;90(6):355-362. doi: 10.3949/ccjm.90a.22052. PMID 37263669
- [Background] Bendtsen L, Zakrzewska JM, Heinskou TB, Hodaie M, Leal PRL, Nurmikko T, Obermann M, Cruccu G, Maarbjerg S. Advances in diagnosis, classification, pathophysiology, and management of trigeminal neuralgia. Lancet Neurol. 2020 Sep;19(9):784-796. doi: 10.1016/S1474-4422(20)30233-7. PMID 32822636
- [Background] Fan X, Fu Z, Ma K, Tao W, Huang B, Guo G, Huang D, Liu G, Song W, Song T, Xiao L, Xia L, Liu Y. Chinese expert consensus on minimally invasive interventional treatment of trigeminal neuralgia. Front Mol Neurosci. 2022 Jul 28;15:953765. doi: 10.3389/fnmol.2022.953765. eCollection 2022. PMID 35966020
- [Background] Abd-Elsayed A, Martens JM, Fiala KJ, Izuogu A. Pulsed Radiofrequency for the Treatment of Trigeminal Neuralgia. Curr Pain Headache Rep. 2022 Dec;26(12):889-894. doi: 10.1007/s11916-022-01092-0. Epub 2022 Nov 15. PMID 36378398
- [Background] Luo F, Meng L, Wang T, Yu X, Shen Y, Ji N. Pulsed radiofrequency treatment for idiopathic trigeminal neuralgia: a retrospective analysis of the causes for ineffective pain relief. Eur J Pain. 2013 Sep;17(8):1189-92. doi: 10.1002/j.1532-2149.2012.00278.x. Epub 2013 Jan 16. PMID 23322665
- [Background] Chua NH, Halim W, Beems T, Vissers KC. Pulsed radiofrequency treatment for trigeminal neuralgia. Anesth Pain Med. 2012 Spring;1(4):257-61. doi: 10.5812/aapm.3493. Epub 2012 Apr 1. PMID 24904811
- [Background] Zipu J, Hao R, Chunmei Z, Lan M, Ying S, Fang L. Long-term Follow-up of Pulsed Radiofrequency Treatment for Trigeminal Neuralgia: Kaplan-Meier Analysis in a Consecutive Series of 149 Patients. Pain Physician. 2021 Dec;24(8):E1263-E1271. PMID 34793653
- [Background] Agarwal A, Rastogi S, Bansal M, Kumar S, Malviya D, Thacker AK. Radiofrequency Treatment of Idiopathic Trigeminal Neuralgia (Conventional vs. Pulsed): A Prospective Randomized Control Study. Anesth Essays Res. 2021 Jan-Mar;15(1):14-19. doi: 10.4103/aer.aer_56_21. Epub 2021 Aug 30. PMID 34667342
- [Background] Everts P, Onishi K, Jayaram P, Lana JF, Mautner K. Platelet-Rich Plasma: New Performance Understandings and Therapeutic Considerations in 2020. Int J Mol Sci. 2020 Oct 21;21(20):7794. doi: 10.3390/ijms21207794. PMID 33096812
- [Background] Gupta S, Paliczak A, Delgado D. Evidence-based indications of platelet-rich plasma therapy. Expert Rev Hematol. 2021 Jan;14(1):97-108. doi: 10.1080/17474086.2021.1860002. Epub 2020 Dec 17. PMID 33275468
- [Background] Hassanien M, Elawamy A, Kamel EZ, Khalifa WA, Abolfadl GM, Roushdy ASI, El Zohne RA, Makarem YS. Perineural Platelet-Rich Plasma for Diabetic Neuropathic Pain, Could It Make a Difference? Pain Med. 2020 Apr 1;21(4):757-765. doi: 10.1093/pm/pnz140. PMID 31298289
- [Background] Zhou Z, Hu X, Yan F, Zhou Y, He R, Ye X, Jiang Z. Observation on the effect of platelet-rich plasma combined with drugs in the treatment of herpes zoster neuralgia. Int J Neurosci. 2024 Jun;134(6):628-634. doi: 10.1080/00207454.2022.2138381. Epub 2022 Nov 2. PMID 36259487
- See also: {Doss2012TrigeminalNT, title={Trigeminal Neuralgia Treatment: A Case Report On Short-Term Follow Up After Ultrasound Guided Autologous Platelet Rich Plasma Injections.}, author={Arockia X Doss}, year={2012} — http://api.semanticscholar.org/CorpusID:79334899